CLINICAL TRIAL: NCT05463770
Title: An Open-Label, Fixed Sequence, Multiple Dose Study of Glucose and Insulin Associated Parameters: SEP-363856 vs Prior Antipsychotic (PA) Standard of Care in Subjects With Schizophrenia Suffering From Metabolic Dysregulation
Brief Title: A Clinical Study That Will Assess the Effect of SEP-363856 and Prior Antipsychotic (PA) Standard of Care on Glucose and Regulation of Insulin in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP361-123
Record Dates: First submitted 2022-07-06; First posted 2022-07-19 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: This is an open-label, fixed sequence, multiple dose design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SEP-363856 (Experimental)
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856, 12.5 mg, 25 mg, and 50 mg tablets. The dose taken at the same time each day, in the evening and in the morning. Multiple tablets may be required to achieve a single dose.

SUMMARY:
A Clinical Study that will look at an investigational medication, SEP-363856 (called "study medication") in patients with schizophrenia and assess whether it changes:

* how the body processes (uses) glucose (blood sugar)
* how much insulin the pancreas can make. Insulin is a hormone that lowers blood sugar levels in the body.

The information from this study will help to understand any effect the study medication may have on how the body uses and stores glucose.

This study is accepting both male and female subjects. It will be held in approximately 6 locations in the United States. Participation could last up to 12 weeks.

DETAILED DESCRIPTION:
This is an open-label, fixed sequence, multiple dose design. Following screening evaluations, subjects will check-in to the clinical research unit. After confirmation of continuation criteria, subjects will undergo an oral glucose tolerance test (oGTT), mixed meal tolerance test (MMTT) and spirulina breath test (GEBT). After these assessments are completed, subjects will have their prior antipsychotic (PA) or any other medication with psychotropic propensity washed out (dependent on their antipsychotic elimination half-life).

Subjects will undergo SEP-363856 titration schedule, followed by the oGTT, MMTT and GEBT tests during the SEP-363856 Stable Dose Period.

Subjects will be stabilized on their prior antipsychotic, discharged from the clinical research unit, and return to the unit for the follow-up visit 7 + 2 days after discharge.

ELIGIBILITY:
Inclusion Criteria: (this list is not all inclusive)

* Male or female subjects between 18 and 65 years of age, inclusive at time of consent.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for a primary diagnosis of schizophrenia as established by clinical interview, using the DSM-5 as a reference and confirmed using the Structured Clinical Interview for DSM-5, Clinical Trials Version [SCID-CT]).
* Subject must have a CGI-S score ≤ 4 (normal to moderately ill) at Screening
* Subject must have a PANSS total score ≤ 80 at Screening and a score of ≤ 4 on the following PANSS items at Screening: P7 (hostility) and G8 (uncooperativeness)
* Subjects' antipsychotic medication at screening must have had no dose change (minor dose adjustments for tolerability purposes are permitted) for at least eight weeks prior to the Screening visit.

Exclusion Criteria: (this list is not all inclusive)

-- Subject has a DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia or intellectual disability (IQ < 70).

* Subject has attempted suicide within 12 months prior to Screening.
* Subject answers "yes" to "Suicidal Ideation" Items 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS at Screening (ie. in the past 1 month) or at any subsequent C-SSRS assessment prior to dosing (ie, since last visit).
* Subject is at risk of harming him/herself or others according to the Investigator's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline (PA) in oGTT derived plasma AUC0-120 min of glucose, insulin, c-peptide in oGTT to stable dose (SEP-363856) period assessment. | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)
Change from baseline (PA) in mixed meal tolerance test (MMTT) derived plasma AUC0-240 min of glucose, insulin, c-peptide and β-cell responsivity index to stable dose (SEP-363856) period assessment. | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)

SECONDARY OUTCOMES:
Change from baseline (PA) in plasma AUC0-240 min and Cmax of acetaminophen levels to stable dose (SEP-363856) period assessment. | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)
Change in Cmax of acetaminophen levels to stable dose (SEP-363856) period assessment. | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)
Change in gastric emptying terminal elimination half-life (T1/2), baseline to stable dose (SEP-363856) period assessment. | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)
Change in kPCD, baseline to stable dose (SEP-363856) period assessment | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)
Change in the Visual Analog Scale (VAS) of fullness, hunger and satiety, baseline - repeat test (PA baseline to SEP-363856 stable dose period assessment) for all time points. | PA Baseline and SEP-363856 Stable Dose Period (up to 48 days)
  Visual Analog Scale (VAS) is on a scale of 0-100, higher represents higher pain intensity (higher score represents worse outcome).
Change in lag time, baseline to stable dose (SEP-363856) period assessment | PA Baseline and SEP-363856 Stalbe Dose Period (up to 48 days)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Catalina Research Institute LLC, Montclair, California
  - CNRI - San Diego LLC, San Diego, California
  - Galiz Research, Hialeah, Florida
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - Pillar Clinical Research, LLC, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com